CLINICAL TRIAL: NCT06595901
Title: Characterizing Mental and Cognitive Health and Physical Activity in the Perioperative Breast Cancer Setting
Brief Title: Mental and Cognitive Health and Physical Activity in the Perioperative Breast Cancer Setting
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 202201163; P50MH122351 (NIH)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Breast Neoplasms; Cancer, Breast; Cancer of the Breast
Keywords: Breast cancer; Physical activity; Prehabilitation; Cognition; Stakeholder needs; Implementation science
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Participants wear ActiGraphs, complete questionnaires via phone call/text message, and participate in interviews remotely on study.
  Interventions: Other: Actigraph; Other: Questionnaires; Other: BrainBaseline application; Other: Semi-structured interviews
- Stakeholders: Semi-structured interviews will be conducted with up to 15 key stakeholders (e.g., nurse coordinators, surgical and medical oncologists, physical therapists) at Siteman Cancer Center.
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Actigraph — Participants will wear an Actigraph hip-worn accelerometer on their non-dominant hip during all waking hours, and on the wrist while sleeping
  Groups: Patients
Other: Questionnaires — * Patient Health Questionnaire Anxiety and Depression Scale30 (PHQ-ADS), a validated composite of anxiety and depressive symptoms.
  * Self-reported cognition will be assessed by the Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog).
  Groups: Patients
Other: BrainBaseline application — Objective measures of cognitive function will include those from the BrainBaseline application, a validated research tool developed by Digital Artefacts to remotely measure domains of cognition
  Groups: Patients
Other: Semi-structured interviews — Semi-structured individual interviews will be conducted with up to 15 healthcare stakeholders and 15-30 patients with breast cancer at any time during the study period, as determined by participant preference.

SUMMARY:
This study evaluates the complex relationships between mental health, cognitive function, and physical activity before surgery in patients with stage I-III breast cancer. Most patients with breast cancer experience declines in their mental health, with up to two-thirds of patients reporting symptoms of depression and anxiety. Cancer-related cognitive decline is even more prevalent; 75% of patients with breast cancer report varying degree of loss in mental acuity throughout their cancer experience. Both mental and cognitive health declines are pervasive, lasting anywhere from 5 years to decades after treatment completion. Not only are these declines detrimental to patients' quality of life, but they also increase the risk of cancer-related mortality. Maintaining sufficient levels of physical activity (PA) is important to both prevent breast cancer and improve health post-diagnosis. PA improves anxiety and depressive symptoms during and after treatment. Early intervention with PA prior to or during cancer treatment, or prehabilitation, can avoid or reduce the severity of treatment-related side effects, hospital length of stay, surgical complications, and care costs. Information gained in this study may help researchers learn more about the right time during treatment for delivering lifestyle programs to improve mental and cognitive health.

ELIGIBILITY:
Eligibility Criteria Patients:

* A physician-confirmed diagnosis of breast cancer (stage I-III)
* Female over the age of 18
* Scheduled to receive curative-intent breast surgery and chemotherapy (neoadjuvant or adjuvant)
* Able to understand and willing to sign an Institutional Review Board (IRB)-approved informed consent document. Given documented mental and cognitive health declines after both neoadjuvant and adjuvant treatment regimens, the investigators are including both patient populations in this exploratory study. Patients of all baseline anxiety, depression, cognitive function, and physical activity levels are eligible to participate.

Eligibility Criteria Stakeholders:

* Healthcare personnel with a staked interest in patient care during chemotherapy, including but not limited to surgical oncologists, medical oncologists, physical and occupational therapists, nurses, patient navigators, dietitians, and exercise physiologists
* Able to understand and willing to sign an IRB-approved informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stages I-III breast cancer at Siteman Cancer Center (SCC) and stakeholders drawn from the surrounding BJC and Washington University healthcare systems.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | Through completion of surgery (estimated to be approximately 12-20 weeks)
  Assessed using an Actigraph hip-worn accelerometer
Change in depression and anxiety | Through completion of surgery (estimated to be approximately 12-20 weeks)
  Assessed using the PHQ-ADS
Change in cognitive function (self-reported) | Through completion of surgery (estimated to be approximately 12-20 weeks)
  Assessed using the FACT-Cog
Change in cognitive function (objective) | Through completion of surgery (estimated to be approximately 12-20 weeks)
  Assessed using the BrainBaseline application

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Salerno, Ph.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
To protect participant privacy, deidentified individual participant data and study protocol will be made available to researchers who provide a methodologically sound proposal for any purpose, immediately following publication
Supporting Information: Study Protocol, SAP
Time Frame: Following publication.
Access Criteria: Proposals should be directed to e.salerno@wustl.edu.

REFERENCES:
- See also: Related Info — http://www.siteman.wustl.edu